CLINICAL TRIAL: NCT06258317
Title: Mesh Fixation Versus Non Fixation in Laparoscopic Inguinal Hernioplasty
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mina Makram George, Principal Investigator, Assiut University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: inguinal hernioplasty
Record Dates: First submitted 2023-12-22; First posted 2024-02-14 (Actual); Last update posted 2024-02-14 (Actual); Status verified 2024-02

CONDITIONS: Laparoscopic; Inguinal Hernia; Hernioplasty
MeSH Terms: conditions — Hernia, Inguinal

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mesh fixation (Experimental): Procedure/Surgery: fixation of conventional polypropylene mesh. This group includes patients with fixation of conventional polypropylene mesh.
  Interventions: Procedure: fixation of conventional polypropylene mesh
- Non-mesh fixation (Experimental): Procedure/Surgery: non-fixation of the mesh. This group includes patients without fixation of the mesh.
  Interventions: Procedure: fixation of conventional polypropylene mesh

INTERVENTIONS:
Procedure: fixation of conventional polypropylene mesh — By fixation of the polyprolene mesh,patients will be divided into two groups:
  Group 1 includes patients with fixation of conventional polypropylene mesh. Group 2 includes patients without fixation of the mesh.

SUMMARY:
Inguinal hernia is one of the most common types of abdominal hernias. Laparoscopic hernioplasty of inguinal hernia is a good alternative to traditional open repairs even in simple unilateral primary inguinal hernia in terms of decrease post operative pain and complications with comparable recurrence rates.Two techniques are described in laparoscopic hernioplasty and have been extensively studied in randomised trials. The totally extraperitoneal (TEP) approach is more widely used than the transabdominal preperitoneal (TAPP) approach.

In this study we will compare between the results of mesh fixation and non fixation as regard operative and postoperative data.

ELIGIBILITY:
Inclusion Criteria:

* Any male or female above 18 years old that has uncomplicated inguinal hernia

Exclusion Criteria:

* Patients with contraindications to use laparoscopy as cardiac or immunocompromised patients.
* Patients who are difficult to follow up.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-02 (Estimated); Primary Completion 2027-02 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Comparing fixation of conventional polypropylene mesh versus non fixation of 3D max mesh (anatomically oriented mesh) in laparoscopic trans-abdominal properitoneal (TAPP) inguinal hernia repair | Baseline
  Comparing fixation of conventional polypropylene mesh versus non fixation of 3D max mesh (anatomically oriented mesh) in laparoscopic transabdominal properitoneal (TAPP) inguinal hernia repair as regard operative and postoperative data.By following-up the patient while admitted post-operatively to check scrotal swelling by examination.After discharge contacting the patient 10 days, 20 days, one month, 2 months, 3 months, 6 months, one year, 2 years to check incidence of recurrence of hernia and return to normal life activities.

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed A Rizk, Principal Investigator — Assiut University

REFERENCES:
- [Background] Lockhart K, Dunn D, Teo S, Ng JY, Dhillon M, Teo E, van Driel ML. Mesh versus non-mesh for inguinal and femoral hernia repair. Cochrane Database Syst Rev. 2018 Sep 13;9(9):CD011517. doi: 10.1002/14651858.CD011517.pub2. PMID 30209805
- [Background] Sun P, Cheng X, Deng S, Hu Q, Sun Y, Zheng Q. Mesh fixation with glue versus suture for chronic pain and recurrence in Lichtenstein inguinal hernioplasty. Cochrane Database Syst Rev. 2017 Feb 7;2(2):CD010814. doi: 10.1002/14651858.CD010814.pub2. PMID 28170080